CLINICAL TRIAL: NCT03091582
Title: Pilot Testing of a Rapid-Onset Psychological Therapy Intervention for Depressed Medical Inpatients
Brief Title: Brief Inpatient Psychotherapy for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Waguih IsHak, Vice Chairman for Education & Research Cedars-Sinai Medical Center, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00046076
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Depression
Keywords: Psychological Therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: After being clearly told that participation in the study will not impact subsequent care at CSMC, the patient agrees to participate, the patient will review and sign the informed consent form. Next, the patient will be randomized to either receive CBT or BA therapy, and scheduled for CBT or BA therapy sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral therapy (Experimental): The Cognitive-Behavioral Therapy (CBT) intervention will focus on catastrophizing and rumination. CBT emphasizes the role of cognitive factors and behavioral factors on affective distress.
  Interventions: Behavioral: Cognitive factors; Behavioral: Behavioral factors
- Behavioral Activation (Experimental): Behavioral Activation is grounded in learning theory and posits that lack of positive/active engagement of the person with his/her environment contributes to an increase in avoidant or passive behaviors and decreased reinforcement. An empirically validated treatment, behavioral activation reduces depressive symptoms and increase engagement of pleasant events.
  Interventions: Behavioral: Increase engagement of pleasant events

INTERVENTIONS:
Behavioral: Cognitive factors — The Cognitive-Behavioral Therapy (CBT) intervention will focus on catastrophizing and rumination. CBT emphasizes the role of cognitive and behavioral factors on affective distress
  Arms: Cognitive behavioral therapy
Behavioral: Behavioral factors — The Cognitive-Behavioral Therapy (CBT) intervention will focus on catastrophizing and rumination. Behavioral factors on affective distress.
  Arms: Cognitive behavioral therapy
Behavioral: Increase engagement of pleasant events — Behavioral Activation is grounded in learning theory and posits that lack of positive/active engagement of the person with his/her environment contributes to an increase in avoidant or passive behaviors and decreased reinforcement. An empirically validated treatment, behavioral activation reduces depressive symptoms and increase engagement of pleasant events.
  Arms: Behavioral Activation

SUMMARY:
The primary objective of the proposed pilot study is to seek to compare the efficacy of two brief psychological therapies during inpatient hospitalization - cognitive behavioral therapy (CBT) versus Behavioral Activation for Medical Inpatients with Depression (BAMID or BA) - for improving depressive symptoms, functioning, and quality of life (QOL). The treatments will consist of four sessions, which will be delivered during hospitalization.

DETAILED DESCRIPTION:
First Visit (after Identification by PHQ Intake Score): If, after being clearly told that participation in the study will not impact subsequent care at CSMC, the patient agrees to participate, the patient will review and sign the informed consent form. Next, the subject will be randomized to either receive CBT or BA therapy, and scheduled for CBT or BA therapy sessions. These sessions will be provided subsequently by an attending psychiatrist or health psychologist in Psychiatry (currently Drs. IsHak, Danovitch, Hedrick, Chaudhry, and Sumner).

Study Visits #'s 2 - 5: Details about the four therapy sessions are listed below. Study Participants will participate in therapy in the hospital room, with no other staff or patients present. Family and friends will not be allowed to be present. If nurses need to enter the room during the therapy session, therapy will be temporarily suspended. The treating clinician will choose a time for therapy that minimizes interruption by examining the patient's schedule and consulting with the attending psychiatrist.

At the end of Visit #5, the study participant will also be offered a referral, by the attending psychiatrist or health psychologist, to a community-based therapist who is not affiliated with CSMC, and if the subject decides to participate, to continue therapy after discharge. The community-based therapist may or may not utilize the same approach utilized during the study. Community-based therapists will be selected among those who are known in the community to the treating psychiatrist/health psychologist, for whom the treating psychiatrist/psychologist can personally vouch. The treating psychiatrist/psychologist may select a community-based therapist whom the patient can afford, or is covered by the patient's insurance. Study participants and therapist will work together to select a community-based provider for use after discharge. The community-based therapy is not part of the research study and, therefore, subjects will be told that seeking this additional therapy is up to the subject and any potential costs related to these sessions will be covered by the subject and/or their insurance company. In the event of early discharge based on medical reasons, the therapy will be concluded and the patient will be referred to the community-based therapist. This will be considered an incomplete delivery of the sessions (early withdrawal).

Treatments Both treatments will consist of four sessions during inpatient hospitalization.

Cognitive Behavioral Therapy (CBT)

1. Session one = Will last 1.5 hours and focus on depression psychoeducation, orient the study participant to brief CBT, treatment goal settings, and identification of maladaptive thoughts and beliefs. Solicit participant feedback and set agenda. Homework includes patient identifying automatic thoughts and core beliefs and associated emotions. Support and encouragement will be provided.
2. Session two = Will last 50 min and will review homework, introduce cognitive strategies to test the accuracy of those beliefs by identifying and modifying negative thoughts and beliefs that give rise to them. Teach and practice identifying ruminative and catastrophizing thoughts. Will also review cognitive distortions and provide support and encouragement. Homework includes participants identifying ruminative and catastrophizing thoughts and challenging those thoughts. Will also teach relaxation techniques (e.g. deep breathing, guided imagery). Support and encouragement will be provided.
3. Session three = Will last 50min and focus on reviewing homework, monitoring moods and activities, planning of exercises to test negative beliefs, and thought records to identify and examine the accuracy of negative automatic thoughts and underlying beliefs. Teach problem-solving skills Provide support and encouragement.
4. Session four = Will last 50 minutes and focus on reviewing and consolidating newly learning cognitive strategies. Practicing. Generate plan for change and provide support and encouragement.

Behavioral Activation for Medical Inpatients with Depression (BAMID or BA)

1. Session one = Will last 1.5 hours of depression psychoeducation (recognition of depression), treatment rationale, assessment of baseline activity level. Identification of factors that contribute to or exacerbate depressive behavior (e.g. withdrawal from friends or family), activity and goal selection, assessment of daily activities and environmental support prior to hospitalization, identification of pleasurable activities in which engaged (could be making a telephone call, journaling, reading, coloring, or if medically stable, having a plaza visit) and homework assignment (reporting a numerical rating of both enjoyment and importance for each activity identified). Provide support and encouragement.
2. Session two = Will last 50 min and include a review of the previous session and completed daily monitoring record forms, an in-depth discussion of life areas and value, and verbal reinforcement of activity engagement. Homework will be to chart progress of activity engagement by duration, frequency, self-reported level of mastery. Provide support and encouragement.
3. Session three =Will last 50 min. Session will include a review of engagement in 3-5 activities considered rewarding and important for values. Discussion of how to continue activities, monitor depressive symptoms and identify rewards for activity engagement. Provide support and encouragement.
4. Session Four = 50 minutes. Will review progress, provide support and encouragement and plan for continued engagement post-discharge. Provide support and encouragement.

Study Visit #6 - Discharge: Before discharge, participants will complete three questionnaires administered by study staff, as follows: 1) a paper version of the PHQ-9 depression inventory, to assess depressive symptoms; 2) the National Institute of Health Patient Reported Outcome Measurement Information System (NIH PROMIS) 10-item Global Health scale, to assess QOL (PROMIS-10); and 3) the World Health Organization Disability Assessment Schedule (WHODAS) 2.0, to assess functioning. These measures will serve as a baseline for comparison with data obtained 90 days later. Participants will also be asked whether they agree to be contacted in 90 days for follow-up assessment; those who agree will be contacted by study staff for Visit #7.

Study Visit #7 - After Discharge: 90 days after the study participant is discharged from the hospital, study staff will contact the subject by phone to inquire about whether they utilized the referral to community-based therapy or not; those who did use the referral will be asked the number of sessions completed over the last 90 days, and the frequency of those sessions. In addition, study staff will also ask whether the subject started antidepressant medication after they left the hospital. If so, they will be asked what the medication and dosage was and how much of the medication they took and (assuming a 30-day dosage), how many pills they have left from the current bottle and when this bottle was prescribed. Any mental health issues that arise during this phone call will be referred to the original attending psychiatrist, or to the community-based therapist if the study participant chose to utilize the referral. Next, the staff member will ask if the study participant is interested in completing study measures over the phone, or on paper. If the subject agrees, the study staff member will administer the same three questionnaires given before discharge over the phone, taking approximately 30 minutes. If the subject prefers to complete these on paper, questionnaires will be mailed by US postal mail along with a self-addressed stamped envelope, and the phone call will end after 5 minutes. These data will be collected and de-identified for analysis.

4 Anticipated Level of Risk:

ELIGIBILITY:
Inclusion Criteria:

* 1) Adults from 18-80; 2) PHQ>12; 3) Medical conditions needing inpatient medical care.

Exclusion Criteria:

* 1) Patients who unable to provide informed consent; 2) Patients deemed in critical medical condition; 3) Conditions that preclude administration of the PHQ for depression screening (e.g., delirium, dementia, acute stroke, loss of consciousness, substance intoxication or withdrawal, agitation, psychotic disorders); 4) Homeless patients, as patient follow-up by mail would be difficult; 5) Meeting criteria for involuntary admission due to imminent danger to self or others, as they are transferred to offsite psychiatric facilities.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Depressive Symptom Severity | 12 weeks
  The PHQ-9 is used to measure depressive symptoms

SECONDARY OUTCOMES:
Functioning | 12 weeks
  WHODAS is used to measure functioning
Overall Health and Quality of life (QOL) | 12 weeks
  NIH-PROMIS-10 is used to measure the overall health and QOL

CONTACTS AND LOCATIONS:
Overall Officials: Waguih W IsHak, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No